CLINICAL TRIAL: NCT06031454
Title: A Open-Label, Two-sequence Phase I Drug-drug Interaction Clinical Study to Investigate the Pharmacokinetics of Leritrelvir With Midazolam, Omeprazole, Rosuvastatin, Verapamil, and Rifampin in Healthy Participants
Brief Title: Drug-durg Interaction of Leritrelvir(RAY1216) With Midazolam, Omeprazole, Rosuvastatin, Verapamil, and Rifampin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: RAY1216-23-05
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — Midazolam; Omeprazole; Rosuvastatin Calcium; Verapamil; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental 1 (Experimental): All participants will receive the following oral doses of study drugs following an overnight fast in the fixed-sequence below:
  Period 1: 1 × 15-mg Midazolam tablet ,1 ×20-mg omeprazole tablet ,1×10-mg rosuvastatin tablet
  Period 2: 6 × 400-mg Leritrelvir tablet+1 × 15-mg Midazolam tablet, 1 ×20-mg omeprazole tablet ,1×10-mg rosuvastatin tablet
  Interventions: Drug: Midazolam; Drug: Omeprazole; Drug: Rosuvastatin; Drug: Leritrelvir
- Experimental 2 (Experimental): All participants will receive the following oral doses of study drugs following an overnight fast in the fixed-sequence below:
  Period 1: 1 × 400-mg Leritrelvir tablet
  Period 2: 5 × 240-mg verapamil tablet+1 × 400-mg Leritrelvir tablet
  Period 3: 8 × 600-mg rifampin capsule +1 × 400-mg Leritrelvir tablet
  Interventions: Drug: Verapamil; Drug: Rifampin; Drug: Leritrelvir

INTERVENTIONS:
Drug: Midazolam — oral
  Arms: Experimental 1
Drug: Omeprazole — oral
  Arms: Experimental 1
Drug: Rosuvastatin — oral
  Arms: Experimental 1
Drug: Verapamil — oral
  Arms: Experimental 2
Drug: Rifampin — oral
  Arms: Experimental 2
Drug: Leritrelvir — oral

SUMMARY:
The drug-drug interaction study had been designed to investigate the effect of Leritrelvir on the pharmacokinetics of Midazolam, Omeprazole, Rosuvastatin and the effect of Verapamil and Rifampin on the pharmacokinetics of Leritrelvir

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥19 to ≤26kg/m2 and total body weight >50 kg(male) or >45kg(female) at screening (calculated as a function of measured height and weight according to the formula, BMI = kg/m2 where m2 is height in meters squared);
2. Ability to understand and willingness to sign a written informed consent form;
3. Normal physical examination,vital signs,12-lead ECG, and clinical laboratory values, or any abnormality that is non-clinically significant.

Exclusion Criteria:

1. Participants with a history of hypersensitivity to study drug(Leritrelvir,Midazolam,Omeprazole,Rosuvastatin, Verapamil, and Rifampin) or any component of study medication;
2. Participants had taken prescription, over-the-counter, herbal, or vitamin products within 14 days prior to screening；
3. Smoking more than 5 cigarettes per day within 3 months prior to screening，or who cannot stop using any tobacco products during the study period;
4. Participants who donated blood/bleeding profusely (>400 mL) 3 months prior to randomization;
5. Those with clinically significant Electrocardiogram(ECG) abnormalities, or QTcF>450ms;
6. Participants who test positive at screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody or Syphilis spirochete-specific antibodies (TPPA);
7. Participants who test positive at screening and/or admission (Day -1) for alcohol abuse.
8. Females who are pregnant, lactating, or likely to become pregnant during the study.
9. History of dysphagia or any gastrointestinal disorder that affect absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - Cmax | 0-72 hours
  Maximum observed plasma concentration
Pharmacokinetic -Area under the curve（AUC） | 0-72 hours
  Area under the curve

SECONDARY OUTCOMES:
Number of participants with adverse events | Day1-Day31
  The safety and tolerability of Leritrelvir alone and in combination with Midazolam, Omeprazole, Rosuvastatin, Verapamil, and Rifampin will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided